CLINICAL TRIAL: NCT03065946
Title: Therapeutic Hypothermia and eArly Waking
Acronym: THAW
Status: Completed | Type: Observational
Sponsor: Mid and South Essex NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: B784
Record Dates: First submitted 2017-02-20; First posted 2017-02-28 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Out of Hospital Cardiac Arrest; Brain Injury
Keywords: Therapeutic hypothermia; Electroencephalogram; Neuron-Specific Enolase; Return of Spontaneous Circulation; S-100B
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Case series: Early wakening
  Interventions: Other: Early wakening

INTERVENTIONS:
Other: Early wakening — By using an intravascular device to administer mild TH for 24 hours, patients can safely have their medically induced coma reversed early at 12 hours, allowing an accurate neurological assessment to be performed

SUMMARY:
Unconscious survivors of cardiac arrest who are treated with intravenous therapeutic hypothermia for 24 hours will be assessed after 12 hours for appropriateness to be woken early and extubated whilst continuing to receive therapeutic hypothermia. Sedation will be reduced/stopped at 12 hours to enable a comprehensive neurological assessment utilising a multimodal approach.

Providing the patient is clinically stable with no adverse neurological signs the patient will be extubated. Patients who remain unconscious will be reviewed 6 hourly for neurological recovery and their suitability to be extubated in line with standard practice.

DETAILED DESCRIPTION:
This study is a single centre, prospective, feasibility and safety study. Consecutively enrolling 50 patients. Subjects will include adult patients who have suffered a cardiac arrest with a return of spontaneous circulation (ROSC).

To qualify, patients must be unconscious and intubated because their initial Glasgow Coma Score (GCS) is <8. Intravenous therapeutic hypothermia (TH) will be established in the cathlab and maintained for 24 hours whilst being cared for in the intensive Care Unit (ICU). IVTM will maintain the patient's core temperature at a target temperature between 32-34 degrees Celsius. After the patient has received 12 hours of TH, sedation will be stopped and the patient will have a comprehensive neurological assessment combining electroencephalogram (EEG), Somatic Sensory Evoked Potential (SSEP) and neurological biomarkers, Neuron Specific Enolase (NSE) and S100b. The EEG, SSEP and biomarkers will be reviewed by an expert in neurophysiology at a core lab off-site. These results will be reviewed retrospectively, therefore will not influence the medical management of the patient.

Patients who are clinically stable and not showing any adverse neurological signs will be extubated after 12 hours. Patients who don't meet the early waking criteria will reassessed every 6 hours for extubation. Those patients who are not suitable to be woken early or remain unconscious after 24 hours will be reassessed as per standard practice for unconscious survivors of cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

* Post cardiac arrest with ROSC
* Planning to receive MTH as part of post-cardiac arrest care

Exclusion Criteria:

* Cardiac arrest caused by trauma, head injury, massive haemorrhage, drug overdose, cerebrovascular accident, drowning, electric shock or hanging.
* Do Not Attempt to Resuscitate (DNAR) orders
* Known terminal illness (e.g. malignancy in the end stages)
* Known or obvious pregnancy
* Known coagulation disorder (except those induced by medication)
* Known oxygen dependency
* The patient has a height of <1.5 meters (4 feet 11 inches)
* The patient has a known hypersensitivity to Buspirone Hydrochloride or Pethidine
* Patient has a known history of severe hepatic or renal impairment, untreated hypothyroidism, Addison's disease, benign prostatic hypertrophy, or urethral stricture that in the opinion of the treating consultant would be incompatible with Pethidine administration
* The patient has an inferior Vena Cava (IVC) filter in place
* The patient has a known, unresolved history of drug use or alcohol dependency, or lacks the ability to comprehend or follow instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiac arrest
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
The number of unconscious survivors following an OHCA, who are admitted to the ICU being treated with MTH who are clinically stable can be safely woken and extubated after 12 hours whilst continuing to receive therapeutic hypothermia. | 12 hours
  Is it safe and feasible to wake patients early whilst receiving therapeutic hypothermia to assess their neurological function?

SECONDARY OUTCOMES:
Reduction in ICU and hospital stay | 24 hours
  Length of ICU and hospital stay
Reduction of Neurological recovery at 12 hours | 24 hours
  Length of time to perform a neurological assessment and intervention
Reduction in the time to perform a CPC assessment | 24 days
  Length of time to perform a Cerebral Performance Category (CPC) assessment
NSE and S100B values during early waking phase | 2 days
  Time of peak NSE and S100B
Composite outcome off all-cause mortality and poor neurological function | 7 days
  Time taken to confirm poor neurological outcome or death
Presence of EEG findings associated with seizures or poor prognosis | 2 days
  Time of identifying abnormal EEG findings associated with seizures or poor prognosis
Presence of SSEP findings associated with poor prognosis | 2 Weeks
  Time of identifying abnormal SSEP findings associated with poor prognosis
Safe to wake unconscious survivors whilst still providing IVTM | 2 Weeks
  Length of time patients are unconscious whilst receiving IVTM

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Keeble, MBBS MD MRCP, Principal Investigator — Basildon and Thurrock University Hospitals NHS FT
Locations (1):
- The Essex Cardiothoracic Centre, Basildon, Essex, United Kingdom

IPD SHARING:
Plan to Share IPD: No